CLINICAL TRIAL: NCT02755844
Title: A Phase I/II Trial to Assess the Safety and Efficacy of Metronomic Cyclophosphamide, Metformin and Olaparib in Recurrent Advanced/Metastatic Endometrial Cancer Patients
Brief Title: Safety and Efficacy of Metronomic Cyclophosphamide, Metformin and Olaparib in Endometrial Cancer Patients
Acronym: ENDOLA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL15_0321
Record Dates: First submitted 2016-04-14; First posted 2016-04-29 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Endometrial Cancer
Keywords: endometrial carcinomas; metronomic cyclophosphamide; metformin; olaparib; dose-escalation study
MeSH Terms: conditions — Endometrial Neoplasms | interventions — olaparib; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib, metformin and metronomic cyclophosphamide (Experimental): Phase 1: Dose escalation scheme: a continual reassessment method (CRM) will be used to guide inclusion of patients in drug dose levels pre-specified based on observations of dose-limiting toxicity.
  Phase 2 (expansion of cohort): once RP2D will be determined, additional patients will be enrolled, in order to obtain preliminary data about efficacy in a 2 stage Simon's design.
  Interventions: Drug: Olaparib; Drug: metformin; Drug: metronomic cyclophosphamide

INTERVENTIONS:
Drug: Olaparib — Olaparib tablet dose will be dose-escalated on 4 dose levels , guided by a continual reassessment method (CRM).
  One cycle will be 28 days (4 weeks) in duration, except for cycle 1 which will be 6 weeks.
Drug: metformin — From week 3 metformin will be gradually escalated from 500 mg/day to 1500 mg/day with weekly 500 mg dose escalation levels
Drug: metronomic cyclophosphamide — from week 2 Metronomic cyclophosphamide will be given continuously on an oral daily basis at 50 mg qd

SUMMARY:
Endometrial cancer ranks 11th in terms of incidence (7275 / year) and mortality (2025 deaths/ year). The 5-year overall survivals of patients at diagnosis with locally advanced and metastatic carcinomas are about 50% and 15% respectively. Beyond first line treatment with platinum-based chemotherapy, there is lack of effective drug in this disease, which explains the poor prognosis of patients.

The prognosis of metastatic endometrial cancer patients is poor, and few drugs have been shown to be effective beyond first chemotherapy line.

Endometrial carcinomas are characterized by frequent alterations of PI3K-AKT-mTor; IGF1R and of DNA repair pathways. Phosphatase and tensin homologue (PTEN)-phosphoinositide 3-kinase (PI3K)-mammalian target of rapamycin (mTor) and DNA repair pathways interact, and inhibition of PI3K-AKT-mTor signaling pathway may alter DNA damage repair.

Metronomic cyclophosphamide regimen may increase the anti-proliferative effects of olaparib because it is an alkylating agent, and it exerts anti-angiogenic effects, with a favorable toxicity profile.

Metformin may increase the anti-proliferative effects of olaparib because it downregulates IGF1R and PI3K-AKT-mTor pathways, with no additive toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Woman older than 18 years and younger than 81 year old
* Patients with histologically and/or cytologically documented endometrial carcinoma (type I or type II), recurrent after platinum-based chemotherapy.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Archival tumor tissue available, or tumor lesion biopsy feasible
* There is no limitation to prior number of therapies
* Patients who have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Patients with adequate bone marrow function

  * Absolute neutrophile count ≥ 1.5 x 10 9 /L
  * Platelet count ≥ 100 x 10 9 /L
  * Haemoglobin ≥ 9 g/dL
* Patients with adequate renal function :

  * Calculated creatinine clearance, using the MDRD formula, according to the standardized IDMS method (http://www.sfndt.org/sn/eservice/calcul/eDFG.htm by ticking IDMS standardized measurement).>= 60 ml/min
* Patients with adequate hepatic function

  *Serum total bilirubin < 1.25 x upper normal limit (UNL) and aspartate aminotransferase (AST)/Alanine Amino transferase (ALT) ≤ 2.5 X UNL (≤ 5 X UNL for patients with liver metastases)
* Patients must have a life expectancy ≥ 16 weeks
* Female patients who are of childbearing potential: evidence of non-childbearing status, practicing practicing two medically acceptable methods of birth control since consent signature during the study and 12 months after the end of treatment
* Patients who gave its written informed consent to participate to the study
* Patients affiliated to a social insurance regime

Exclusion Criteria:

* Illness, incompatible with metformin treatment, in particular those associated with a risk of hypoperfusion or hypoxia (not limited to): acute or chronic renal failure (creatinine clearance < 60 ml/min, using the MDRD formula according to the standardized IDMS method); lactic ketoacidosis; septic shock; congestive heart failure; respiratory distress; liver failure; chronic alcoholism; uncontrolled seizures; age > 80 years; allergy/hypersensitivity to metformin.
* Previous treatment with cyclophosphamide; or allergy/hypersensitivity to cyclophosphamide or one of its excipients or one of its metabolits.
* Illness incompatible with cyclophosphamide treatment: pre-existing hemorrhagic cystitis and urinary tract obstruction
* Any previous treatment with a poly-adenosine diphosphate ribose (ADP) ribose polymerase (PARP) inhibitor, including olaparib.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment. The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Concomitant use of known CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin boceprevir, telaprevir and nelfinavir and inducers such phenobarbital, phenytoin, carbamazepine, rifampicin.
* Persistent toxicities (>=CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
* Treatment with other investigational agents.
* Bowel occlusive syndrome or other gastro-intestinal disorder that does not allow oral medication such as malabsorption.
* Female patients who are pregnant or lactating, Active infection to HIV, hepatitis B or C, or have other forms of hepatitis or cirrhosis.
* Symptomatic uncontrolled brain metastases. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
* Major surgery within 14 days of starting study treatment
* Patients must have recovered from any effects of any major surgery.
* Resting ECG with corrected QT interval (QTc) > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Concomitant treatment with vitamin K antagonists
* Patients under guardianship.

A diabetic patient may be included in the study. In that case:

- If the patient is treated with metformin: Keep metformin at the usual dosage. There will be no prescription or dispensation in the study.

- If the patient is being treated with another medicine (ex Stagid): Take the advice of a diabetologist or the referring physician for the patient's diabetes for the continuation of the same treatment and the addition of metformin to 500 mg/day.

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 trial (RP2D) dose of olaparib combined to metronomic cyclophosphamide and metformin | through the 6th week of treatment (cycle 1)

SECONDARY OUTCOMES:
Efficacy of olaparib combined to metronomic cyclophosphamide and metformin | at 10 weeks
  non-progression rate at 10 weeks, calculated as the combination of stable disease, partial response and complete response defined according to RECIST v.1.1
Number of patients with adverse events relative to the study treatment olaparib combined to metronomic cyclophosphamide and metformin | through treatment completion (a median of 12 months)
  All adverse events relative to the study treatment will be recorded (NCI- Common Terminology for Adverse Events (CTAE) v.4 criteria) during the treatment.
Pharmacodynamic effects of the 3 drugs on circulating tumor DNA (ctDNA), | through treatment completion (a median of 12 months)
  The kinetics of circulating tumor DNA (ctDNA), serially measured will be assessed using population kinetic approach and mathematical modeling
Pharmacodynamic effects of the 3 drugs on circulating Insulin Growth Factor (IGF-1) | through treatment completion (a median of 12 months)
  The kinetics of Insulin Growth Factor (IGF-1) values serially measured will be assessed using population kinetic approach and mathematical modeling
Pharmacodynamic effects of the 3 drugs on circulating (Cancer Antigen) CA-125 values | through treatment completion (a median of 12 months)
  The kinetics of (Cancer Antigen) CA-125 values serially measured will be assessed using population kinetic approach and mathematical modeling

CONTACTS AND LOCATIONS:
Overall Officials: Benoit YOU, Doctor, Principal Investigator — Hospices Civils de Lyon
Locations (6):
- France (6):
  - Service d'Oncologie Médicale, Centre François Baclesse, Caen
  - Département de Cancérologie Cervico-Faciale et Thoracique, Centre Oscar Lambret, Lille
  - Département d'Oncologie Médicale, Centre Antoine Lacassagne, Nice
  - Service d'Oncologie Médicale, Institut Curie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Comité Gynécologique, Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piffoux M, Leary A, Follana P, Abdeddaim C, Joly F, Bin S, Bonjour M, Boulai A, Callens C, Villeneuve L, Alexandre M, Schwiertz V, Freyer G, Rodrigues M, You B. Olaparib combined to metronomic cyclophosphamide and metformin in women with recurrent advanced/metastatic endometrial cancer: the ENDOLA phase I/II trial. Nat Commun. 2025 Feb 20;16(1):1821. doi: 10.1038/s41467-025-56914-7. PMID 39979249